CLINICAL TRIAL: NCT00088699
Title: Investigation of the Rapid (Next Day) Antidepressant Effects of an NMDA Antagonist
Brief Title: Rapid Antidepressant Effects of Ketamine in Major Depression
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 040222; 04-M-0222
Record Dates: First submitted 2004-07-30; First posted 2004-08-02 (Estimated); Results first posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2017-07-31

CONDITIONS: Depression; Mood Disorders; Major Depresssion
Keywords: Depression; NMDA Antagonist; Treatment Resistant; Glutamatergic System; Major Depression
MeSH Terms: conditions — Depression; Mood Disorders; Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine, Then Placebo (Experimental): Ketamine and placebo infusions were administered two weeks apart, with Ketamine's dose being 0.5 mg/kg.
  Interventions: Drug: Ketamine; Drug: Placebo
- Placebo, Then Ketamine (Experimental): Placebo and Ketamine infusions were administered two weeks apart, with Ketamine's dose being 0.5 mg/kg
  Interventions: Drug: Ketamine; Drug: Placebo

INTERVENTIONS:
Drug: Ketamine
Drug: Placebo

SUMMARY:
Depressive disorders may be severe, chronic and often life-threatening illnesses. Impairment in physical and social functioning resulting from depression can be just as severe as other chronic medical illnesses. Recent preclinical and clinical studies suggest that the glutamatergic system is involved in the mechanism of action of antidepressants.

This study examines whether ketamine can cause a rapid-next day antidepressant effect in patients with Major Depressive Disorder.

This study was designed to address the questions:

Does the NMDA antagonist ketamine produce rapid antidepressant effects in patients with treatment-resistant major depression? What are the neurobiological correlates of antidepressant response (examining multi-modal MRI, MEG, polysomnography and serum markers) Patients, ages 18 to 65 years with treatment-resistant major (unipolar) depression will in a double-blind crossover study receive either intravenous ketamine or saline solution.

DETAILED DESCRIPTION:
This study will test whether a single dose of ketamine - a drug that blocks a brain receptor called NMDA - can cause a rapid (next day) antidepressant effect in patients with major depression. Several medications are effective for treating depression; however, they take weeks or months to achieve their full effects. A more rapidly acting antidepressant would have a significant impact on the treatment of depression. In a previous study, ketamine produced a rapid antidepressant effect within hours, but the effect lasted less than 1 week. Understanding how ketamine works may lead to a better understanding of the causes of depression and the design of a longer lasting rapidly acting antidepressant.

Patients between 18 and 65 years of age who are currently experiencing an episode of major depression of at least 4 weeks duration and have not responded to two treatment trials may be eligible for this study. Candidates are screened with a medical and psychiatric history, physical examination, and blood and urine tests.

Participants undergo the following tests and procedures:

Medication tapering: Patients who are taking medications for depression are tapered off the drugs over a 1- to 2-week period.

Ketamine/placebo trial: Patients are given a single dose of either ketamine or placebo (an inactive substance), administered intravenously (through a vein) over 40 minutes. After 7 days, patients are given another dose of study drug in crossover fashion; that is, those who previously took ketamine are switched to receive placebo, and those who took placebo are switched to ketamine. Oximetry (measurement of blood oxygen), pulse, and blood pressure are measured continuously for 1 hour before and 4 hours after each ketamine or placebo dose to monitor safety.

Interviews and rating scales: Patients complete a series of psychiatric rating scales to assess the effects of the study drug on mood and thinking. The rating scales are repeated up to 18 times during the study, with each time taking about 15 to 20 minutes.

Physical examination and laboratory tests: Patients have a physical examination, blood tests, weight measure, and electrocardiogram (ECG) at the beginning and end of the study. They will also have multi-modal MRI, MEG, polysomnography and serum marker studies.

The primary endpoint will be the change in clinical ratings of depression. Secondary endpoints will examine neurobiological correlates (i.e., multi-modal MRI, MEG, polysomnography and serum markers) of antidepressant response to ketamine (compared to placebo).

ELIGIBILITY:
* INCLUSION CRITERIA:

General patient inclusion criteria

1. Male or female subjects, 18 to 65 years of age.
2. Each subject must have a level of understanding sufficient to agree to all required tests and examinations and sign an informed consent document.
3. Subjects must fulfill DSM-IV criteria for Major Depressive Disorder (MDD) without psychotic features, based on clinical assessment and confirmed by a structured diagnostic interview, SCID-P.
4. Subjects must have an initial score of at least 20 on the MADRS at screen and at baseline of study phase I.
5. Subjects must have failed to respond in the past to an adequate dose and duration of at least one antidepressant (SSRI, bupropion, or venlafaxine) during a depressive episode
6. Current depressive episode of at least 4 weeks duration.

Additional inclusion criteria for substudy 4 (patients with MDD)

1. Age of onset less than 40 years of age.
2. Subjects with MDD must fulfill DSM-IV criteria for Major Depression single episode or recurrent without psychotic features based on clinical assessment and confirmed by a structured diagnostic interview (SCID-P).
3. A failed adequate trial of ECT would count as an adequate antidepressant trial.
4. In women of childbearing age, a negative pregnancy test within 24 hours of MRI.

Inclusion criteria for healthy control subjects (Substudy 4 only)

1. Age 18-65 years.
2. Written informed consent completed.

EXCLUSION CRITERIA:

General patient exclusion criteria

1. Current or past diagnosis of Schizophrenia or any other psychotic disorder as defined in the DSM-IV.
2. Subjects with a history of DSM-IV drug or alcohol dependency or abuse (except for nicotine or caffeine) within the preceding 3 months.
3. Female subjects who are either pregnant or nursing.
4. Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
5. Subjects with uncorrected hypothyroidism or hyperthyroidism.
6. Subjects with one or more seizures without a clear and resolved etiology.
7. Treatment with a reversible MAOI within 4 weeks prior to study phase I.
8. Treatment with fluoxetine within 5 weeks prior to study phase I.
9. Treatment with any other concomitant medication not allowed (Appendix A for Substudy 2; Appendix G for Substudy 4) 14 days prior to study phase I.
10. No structured psychotherapy will be permitted during the study.
11. Current NIMH employee/staff or their immediate family member.

Additional Exclusion Criteria for substudy 2 (patients with MDD)

1. Previous treatment with ketamine or hypersensitivity to amantadine.

Additional Exclusion Criteria for Substudy 4 (patients with MDD)

1. Subjects who currently are using drugs (except for caffeine or nicotine), must not have used illicit substances in the 2 weeks prior to screen and must have a negative alcohol and drug urine test (except for prescribed benzodiazepines) urine test at screening.
2. Presence of any medical illness likely to alter brain morphology and/or physiology (e.g., hypertension, diabetes) even if controlled by medications.
3. Clinically significant abnormal laboratory tests.
4. For imaging procedures, Presence of metallic (ferromagnetic) implants (e.g, heart pacemaker, aneurysm clip).
5. Subjects who, in the investigator's judgment, pose a current serious suicidal or homicidal risk, or who have a MADRS item 10 score of >4.

Exclusion Criteria for healthy control subjects (Substudy 4 only)

1. Current or past Axis I diagnosis
2. Presence of metallic (ferromagnetic) implants (e.g., heart pacemaker, aneurysm clips).
3. Presence of medical illness likely to alter brain morphology and/or physiology (e.g., hypertension, diabetes) even if controlled by medications.
4. Treatment with any of the exclusionary medications detailed in Appendix G 14 days prior to Phase 1 of the Substudy 4.
5. Current or past alcohol or substance abuse or dependence diagnosis (except for nicotine or caffeine).
6. Presence of psychiatric disorders in first-degree relatives.
7. Female subjects who are either pregnant or nursing.

7.8.Current NIMH employee/staff or their immediate family member.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2004-07-26; Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Zarate, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Result] Nugent AC, Ballard ED, Gould TD, Park LT, Moaddel R, Brutsche NE, Zarate CA Jr. Ketamine has distinct electrophysiological and behavioral effects in depressed and healthy subjects. Mol Psychiatry. 2019 Jul;24(7):1040-1052. doi: 10.1038/s41380-018-0028-2. Epub 2018 Feb 27. PMID 29487402
- [Result] Evans JW, Lally N, An L, Li N, Nugent AC, Banerjee D, Snider SL, Shen J, Roiser JP, Zarate CA Jr. 7T 1H-MRS in major depressive disorder: a Ketamine Treatment Study. Neuropsychopharmacology. 2018 Aug;43(9):1908-1914. doi: 10.1038/s41386-018-0057-1. Epub 2018 Apr 5. PMID 29748628
- [Result] Gilbert JR, Yarrington JS, Wills KE, Nugent AC, Zarate CA. Glutamatergic Signaling Drives Ketamine-Mediated Response in Depression: Evidence from Dynamic Causal Modeling. Int J Neuropsychopharmacol. 2018 Aug 1;21(8):740-747. doi: 10.1093/ijnp/pyy041. PMID 29668918
- [Result] Evans JW, Szczepanik J, Brutsche N, Park LT, Nugent AC, Zarate CA Jr. Default Mode Connectivity in Major Depressive Disorder Measured Up to 10 Days After Ketamine Administration. Biol Psychiatry. 2018 Oct 15;84(8):582-590. doi: 10.1016/j.biopsych.2018.01.027. Epub 2018 Feb 15. PMID 29580569
- [Result] Nugent AC, Zarate CA Jr. Using Neuroimaging to Decipher the Mechanism of Action of Ketamine: A Pathway to Novel Therapeutics? Biol Psychiatry Cogn Neurosci Neuroimaging. 2017 Oct;2(7):549-551. doi: 10.1016/j.bpsc.2017.08.006. Epub 2017 Oct 5. No abstract available. PMID 29560906
- [Result] Kadriu B, Gold PW, Luckenbaugh DA, Lener MS, Ballard ED, Niciu MJ, Henter ID, Park LT, De Sousa RT, Yuan P, Machado-Vieira R, Zarate CA. Acute ketamine administration corrects abnormal inflammatory bone markers in major depressive disorder. Mol Psychiatry. 2018 Jul;23(7):1626-1631. doi: 10.1038/mp.2017.109. Epub 2017 May 30. PMID 28555075
- [Derived] Kheirkhah M, Hejazi NS, Nugent AC, Gilbert JR, Leistritz L, Walter M, Duncan WC Jr, Goldman D, Zarate CA Jr. Exploring the link between waking gamma and sleep delta power in healthy volunteers and individuals with treatment-resistant depression. J Affect Disord. 2025 Sep 15;385:119448. doi: 10.1016/j.jad.2025.119448. Epub 2025 May 19. PMID 40398609
- [Derived] Kheirkhah M, Duncan WC Jr, Yuan Q, Wang PR, Jamalabadi H, Leistritz L, Walter M, Goldman D, Zarate CA Jr, Hejazi NS. REM density predicts rapid antidepressant response to ketamine in individuals with treatment-resistant depression. Neuropsychopharmacology. 2025 May;50(6):941-946. doi: 10.1038/s41386-025-02066-7. Epub 2025 Feb 15. PMID 39955416
- [Derived] Ballard ED, Greenstein D, Reiss PT, Crainiceanu CM, Cui E, Duncan WC Jr, Hejazi NS, Zarate CA Jr. Functional changes in sleep-related arousal after ketamine administration in individuals with treatment-resistant depression. Transl Psychiatry. 2024 Jun 4;14(1):238. doi: 10.1038/s41398-024-02956-2. PMID 38834540
- [Derived] Alexander L, Hawkins PCT, Evans JW, Mehta MA, Zarate CA Jr. Preliminary evidence that ketamine alters anterior cingulate resting-state functional connectivity in depressed individuals. Transl Psychiatry. 2023 Dec 1;13(1):371. doi: 10.1038/s41398-023-02674-1. PMID 38040678
- [Derived] Punturieri C, Duncan WC Jr, Greenstein D, Shandler G, Zarate CA Jr, Evans JW. An exploration of actigraphy in the context of ketamine and treatment-resistant depression. Int J Methods Psychiatr Res. 2023 Sep 5;33(1):e1984. doi: 10.1002/mpr.1984. Online ahead of print. PMID 37668277
- [Derived] Quintanilla B, Medeiros GC, Greenstein D, Yuan P, Johnston JN, Park LT, Goes FS, Gould TD, Zarate CA Jr. kappa-Opioid Receptor Plasma Levels Are Associated With Sex and Diagnosis of Major Depressive Disorder But Not Response to Ketamine. J Clin Psychopharmacol. 2023 Mar-Apr 01;43(2):89-96. doi: 10.1097/JCP.0000000000001663. PMID 36821406
- [Derived] Hejazi NS, Farmer CA, Oppenheimer M, Falodun TB, Park LT, Duncan WC Jr, Zarate CA Jr. The relationship between the HDRS insomnia items and polysomnographic (PSG) measures in individuals with treatment-resistant depression. J Psychiatr Res. 2022 Apr;148:27-33. doi: 10.1016/j.jpsychires.2022.01.022. Epub 2022 Jan 11. PMID 35092868
- [Derived] Dean RL, Marquardt T, Hurducas C, Spyridi S, Barnes A, Smith R, Cowen PJ, McShane R, Hawton K, Malhi GS, Geddes J, Cipriani A. Ketamine and other glutamate receptor modulators for depression in adults with bipolar disorder. Cochrane Database Syst Rev. 2021 Oct 8;10(10):CD011611. doi: 10.1002/14651858.CD011611.pub3. PMID 34623633
- [Derived] Gilbert JR, Galiano CS, Nugent AC, Zarate CA. Ketamine and Attentional Bias Toward Emotional Faces: Dynamic Causal Modeling of Magnetoencephalographic Connectivity in Treatment-Resistant Depression. Front Psychiatry. 2021 Jun 18;12:673159. doi: 10.3389/fpsyt.2021.673159. eCollection 2021. PMID 34220581
- [Derived] Acevedo-Diaz EE, Greenwald M, Cavanaugh GW, Greenstein DK, Kraus C, Kadriu B, Zarate CA Jr, Park LT. Reply to: "Letter to the Editor: Are ketamine-induced subjective bodily experiences associated with antidepressant effects? A sensation of floating and a sensation of Lightnessare not the same - A comment on Acevedo-Diaz et al." (Jpsychiatrres-D-21-00121). J Psychiatr Res. 2021 May;137:409-410. doi: 10.1016/j.jpsychires.2021.03.018. Epub 2021 Mar 16. No abstract available. PMID 33773443
- [Derived] Lundin NB, Sepe-Forrest L, Gilbert JR, Carver FW, Furey ML, Zarate CA Jr, Nugent AC. Ketamine Alters Electrophysiological Responses to Emotional Faces in Major Depressive Disorder. J Affect Disord. 2021 Jan 15;279:239-249. doi: 10.1016/j.jad.2020.10.007. Epub 2020 Oct 7. PMID 33074143
- [Derived] Mkrtchian A, Evans JW, Kraus C, Yuan P, Kadriu B, Nugent AC, Roiser JP, Zarate CA Jr. Ketamine modulates fronto-striatal circuitry in depressed and healthy individuals. Mol Psychiatry. 2021 Jul;26(7):3292-3301. doi: 10.1038/s41380-020-00878-1. Epub 2020 Sep 14. PMID 32929215
- [Derived] Nugent AC, Ballard ED, Gilbert JR, Tewarie PK, Brookes MJ, Zarate CA Jr. Multilayer MEG functional connectivity as a potential marker for suicidal thoughts in major depressive disorder. Neuroimage Clin. 2020;28:102378. doi: 10.1016/j.nicl.2020.102378. Epub 2020 Aug 8. PMID 32836087
- [Derived] Kraus C, Mkrtchian A, Kadriu B, Nugent AC, Zarate CA Jr, Evans JW. Evaluating global brain connectivity as an imaging marker for depression: influence of preprocessing strategies and placebo-controlled ketamine treatment. Neuropsychopharmacology. 2020 May;45(6):982-989. doi: 10.1038/s41386-020-0624-0. Epub 2020 Jan 29. PMID 31995812
- [Derived] Gilbert JR, Ballard ED, Galiano CS, Nugent AC, Zarate CA Jr. Magnetoencephalographic Correlates of Suicidal Ideation in Major Depression. Biol Psychiatry Cogn Neurosci Neuroimaging. 2020 Mar;5(3):354-363. doi: 10.1016/j.bpsc.2019.11.011. Epub 2019 Dec 3. PMID 31928949
- [Derived] Acevedo-Diaz EE, Cavanaugh GW, Greenstein D, Kraus C, Kadriu B, Zarate CA, Park LT. Comprehensive assessment of side effects associated with a single dose of ketamine in treatment-resistant depression. J Affect Disord. 2020 Feb 15;263:568-575. doi: 10.1016/j.jad.2019.11.028. Epub 2019 Nov 10. PMID 31791675
- [Derived] Kadriu B, Farmer CA, Yuan P, Park LT, Deng ZD, Moaddel R, Henter ID, Shovestul B, Ballard ED, Kraus C, Gold PW, Machado-Vieira R, Zarate CA Jr. The kynurenine pathway and bipolar disorder: intersection of the monoaminergic and glutamatergic systems and immune response. Mol Psychiatry. 2021 Aug;26(8):4085-4095. doi: 10.1038/s41380-019-0589-8. Epub 2019 Nov 15. PMID 31732715
- [Derived] Reed JL, Nugent AC, Furey ML, Szczepanik JE, Evans JW, Zarate CA Jr. Effects of Ketamine on Brain Activity During Emotional Processing: Differential Findings in Depressed Versus Healthy Control Participants. Biol Psychiatry Cogn Neurosci Neuroimaging. 2019 Jul;4(7):610-618. doi: 10.1016/j.bpsc.2019.01.005. Epub 2019 Jan 25. PMID 30826253
- [Derived] Ballard ED, Reed JL, Szczepanik J, Evans JW, Yarrington JS, Dickstein DP, Nock MK, Nugent AC, Zarate CA Jr. Functional Imaging of the Implicit Association of the Self With Life and Death. Suicide Life Threat Behav. 2019 Dec;49(6):1600-1608. doi: 10.1111/sltb.12543. Epub 2019 Feb 13. PMID 30761601
- [Derived] Nugent AC, Wills KE, Gilbert JR, Zarate CA Jr. Synaptic potentiation and rapid antidepressant response to ketamine in treatment-resistant major depression: A replication study. Psychiatry Res Neuroimaging. 2019 Jan 30;283:64-66. doi: 10.1016/j.pscychresns.2018.09.001. Epub 2018 Sep 12. PMID 30551012
- [Derived] Ballard ED, Yarrington JS, Farmer CA, Richards E, Machado-Vieira R, Kadriu B, Niciu MJ, Yuan P, Park L, Zarate CA Jr. Characterizing the course of suicidal ideation response to ketamine. J Affect Disord. 2018 Dec 1;241:86-93. doi: 10.1016/j.jad.2018.07.077. Epub 2018 Jul 30. PMID 30099268
- [Derived] Reed JL, Nugent AC, Furey ML, Szczepanik JE, Evans JW, Zarate CA Jr. Ketamine normalizes brain activity during emotionally valenced attentional processing in depression. Neuroimage Clin. 2018 Jul 5;20:92-101. doi: 10.1016/j.nicl.2018.07.006. eCollection 2018. PMID 30094160
- [Derived] Ballard ED, Yarrington JS, Farmer CA, Lener MS, Kadriu B, Lally N, Williams D, Machado-Vieira R, Niciu MJ, Park L, Zarate CA Jr. Parsing the heterogeneity of depression: An exploratory factor analysis across commonly used depression rating scales. J Affect Disord. 2018 Apr 15;231:51-57. doi: 10.1016/j.jad.2018.01.027. Epub 2018 Feb 5. PMID 29448238
- [Derived] Duncan WC Jr, Slonena E, Hejazi NS, Brutsche N, Yu KC, Park L, Ballard ED, Zarate CA Jr. Motor-Activity Markers of Circadian Timekeeping Are Related to Ketamine's Rapid Antidepressant Properties. Biol Psychiatry. 2017 Sep 1;82(5):361-369. doi: 10.1016/j.biopsych.2017.03.011. Epub 2017 Mar 28. PMID 28457485
- [Derived] Vande Voort JL, Ballard ED, Luckenbaugh DA, Bernert RA, Richards EM, Niciu MJ, Park LT, Machado-Vieira R, Duncan WC Jr, Zarate CA Jr. Antisuicidal Response Following Ketamine Infusion Is Associated With Decreased Nighttime Wakefulness in Major Depressive Disorder and Bipolar Disorder. J Clin Psychiatry. 2017 Sep/Oct;78(8):1068-1074. doi: 10.4088/JCP.15m10440. PMID 27929610
- [Derived] Lepow L, Luckenbaugh DA, Park L, Henter ID, Zarate CA Jr. Case series: Antidepressant effects of low-affinity and low-trapping NMDA receptor antagonists did not predict response to ketamine in seven subjects. J Psychiatr Res. 2017 Mar;86:55-57. doi: 10.1016/j.jpsychires.2016.10.023. Epub 2016 Nov 22. No abstract available. PMID 27914292
- [Derived] Pennybaker SJ, Niciu MJ, Luckenbaugh DA, Zarate CA. Symptomatology and predictors of antidepressant efficacy in extended responders to a single ketamine infusion. J Affect Disord. 2017 Jan 15;208:560-566. doi: 10.1016/j.jad.2016.10.026. Epub 2016 Oct 26. PMID 27839782
- [Derived] Bernert RA, Luckenbaugh DA, Duncan WC, Iwata NG, Ballard ED, Zarate CA. Sleep architecture parameters as a putative biomarker of suicidal ideation in treatment-resistant depression. J Affect Disord. 2017 Jan 15;208:309-315. doi: 10.1016/j.jad.2016.08.050. Epub 2016 Oct 14. PMID 27810712
- [Derived] Park M, Newman LE, Gold PW, Luckenbaugh DA, Yuan P, Machado-Vieira R, Zarate CA Jr. Change in cytokine levels is not associated with rapid antidepressant response to ketamine in treatment-resistant depression. J Psychiatr Res. 2017 Jan;84:113-118. doi: 10.1016/j.jpsychires.2016.09.025. Epub 2016 Sep 30. PMID 27718369
- [Derived] Berg HE, Ballard ED, Luckenbaugh DA, Nugent AC, Ionescu DF, Zarate CA Jr. Recognition of emotional facial expressions in anxious and nonanxious depression. Compr Psychiatry. 2016 Oct;70:1-8. doi: 10.1016/j.comppsych.2016.06.007. Epub 2016 Jun 14. PMID 27624417
- [Derived] Ballard ED, Vande Voort JL, Luckenbaugh DA, Machado-Vieira R, Tohen M, Zarate CA. Acute risk factors for suicide attempts and death: prospective findings from the STEP-BD study. Bipolar Disord. 2016 Jun;18(4):363-72. doi: 10.1111/bdi.12397. Epub 2016 May 27. PMID 27233466
- [Derived] Ballard ED, Luckenbaugh DA, Richards EM, Walls TL, Brutsche NE, Ameli R, Niciu MJ, Vande Voort JL, Zarate CA Jr. Assessing measures of suicidal ideation in clinical trials with a rapid-acting antidepressant. J Psychiatr Res. 2015 Sep;68:68-73. doi: 10.1016/j.jpsychires.2015.06.003. Epub 2015 Jun 16. PMID 26228403
- [Derived] Luckenbaugh DA, Ameli R, Brutsche NE, Zarate CA Jr. Rating depression over brief time intervals with the Hamilton Depression Rating Scale: standard vs. abbreviated scales. J Psychiatr Res. 2015 Feb;61:40-5. doi: 10.1016/j.jpsychires.2014.12.015. Epub 2014 Dec 27. PMID 25592045
- [Derived] Ortiz R, Niciu MJ, Lukkahati N, Saligan LN, Nugent AC, Luckenbaugh DA, Machado-Vieira R, Zarate CA Jr. Shank3 as a potential biomarker of antidepressant response to ketamine and its neural correlates in bipolar depression. J Affect Disord. 2015 Feb 1;172:307-11. doi: 10.1016/j.jad.2014.09.015. Epub 2014 Oct 16. PMID 25451430
- [Derived] Ionescu DF, Luckenbaugh DA, Niciu MJ, Richards EM, Zarate CA Jr. A single infusion of ketamine improves depression scores in patients with anxious bipolar depression. Bipolar Disord. 2015 Jun;17(4):438-43. doi: 10.1111/bdi.12277. Epub 2014 Nov 14. PMID 25400146
- [Derived] Ionescu DF, Luckenbaugh DA, Niciu MJ, Richards EM, Slonena EE, Vande Voort JL, Brutsche NE, Zarate CA Jr. Effect of baseline anxious depression on initial and sustained antidepressant response to ketamine. J Clin Psychiatry. 2014 Sep;75(9):e932-8. doi: 10.4088/JCP.14m09049. PMID 25295436
- [Derived] Ballard ED, Ionescu DF, Vande Voort JL, Niciu MJ, Richards EM, Luckenbaugh DA, Brutsche NE, Ameli R, Furey ML, Zarate CA Jr. Improvement in suicidal ideation after ketamine infusion: relationship to reductions in depression and anxiety. J Psychiatr Res. 2014 Nov;58:161-6. doi: 10.1016/j.jpsychires.2014.07.027. Epub 2014 Aug 12. PMID 25169854
- [Derived] Cornwell BR, Salvadore G, Furey M, Marquardt CA, Brutsche NE, Grillon C, Zarate CA Jr. Synaptic potentiation is critical for rapid antidepressant response to ketamine in treatment-resistant major depression. Biol Psychiatry. 2012 Oct 1;72(7):555-61. doi: 10.1016/j.biopsych.2012.03.029. Epub 2012 Apr 21. PMID 22521148
- [Derived] Zarate CA Jr, Brutsche NE, Ibrahim L, Franco-Chaves J, Diazgranados N, Cravchik A, Selter J, Marquardt CA, Liberty V, Luckenbaugh DA. Replication of ketamine's antidepressant efficacy in bipolar depression: a randomized controlled add-on trial. Biol Psychiatry. 2012 Jun 1;71(11):939-46. doi: 10.1016/j.biopsych.2011.12.010. Epub 2012 Jan 31. PMID 22297150
- [Derived] Diazgranados N, Ibrahim L, Brutsche NE, Newberg A, Kronstein P, Khalife S, Kammerer WA, Quezado Z, Luckenbaugh DA, Salvadore G, Machado-Vieira R, Manji HK, Zarate CA Jr. A randomized add-on trial of an N-methyl-D-aspartate antagonist in treatment-resistant bipolar depression. Arch Gen Psychiatry. 2010 Aug;67(8):793-802. doi: 10.1001/archgenpsychiatry.2010.90. PMID 20679587
- [Derived] DiazGranados N, Ibrahim LA, Brutsche NE, Ameli R, Henter ID, Luckenbaugh DA, Machado-Vieira R, Zarate CA Jr. Rapid resolution of suicidal ideation after a single infusion of an N-methyl-D-aspartate antagonist in patients with treatment-resistant major depressive disorder. J Clin Psychiatry. 2010 Dec;71(12):1605-11. doi: 10.4088/JCP.09m05327blu. Epub 2010 Jul 13. PMID 20673547
- [Derived] Machado-Vieira R, Yuan P, Brutsche N, DiazGranados N, Luckenbaugh D, Manji HK, Zarate CA Jr. Brain-derived neurotrophic factor and initial antidepressant response to an N-methyl-D-aspartate antagonist. J Clin Psychiatry. 2009 Dec;70(12):1662-6. doi: 10.4088/JCP.08m04659. Epub 2009 Sep 8. PMID 19744406
- [Derived] Phelps LE, Brutsche N, Moral JR, Luckenbaugh DA, Manji HK, Zarate CA Jr. Family history of alcohol dependence and initial antidepressant response to an N-methyl-D-aspartate antagonist. Biol Psychiatry. 2009 Jan 15;65(2):181-4. doi: 10.1016/j.biopsych.2008.09.029. Epub 2008 Nov 8. PMID 18996507
- [Derived] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061

RESULTS

PARTICIPANT FLOW:
Groups:
- MDD: Ketamine, Then Placebo: Ketamine and placebo infusions were administered two weeks apart, with Ketamine's dose being 0.5 mg/kg.
- MDD: Placebo, Then Ketamine; Healthy Volunteers: Ketamine, Then Placebo; Healthy Volunteers:Placebo, Then Ketamine: Placebo and Ketamine infusions were administered two weeks apart, with Ketamine's dose being 0.5 mg/kg
Period: Infusion 1
Arm/Group | MDD: Ketamine, Then Placebo | MDD: Placebo, Then Ketamine | Healthy Volunteers: Ketamine, Then Placebo | Healthy Volunteers:Placebo, Then Ketamine
Started | 23 | 19 | 13 | 12
Completed | 22 | 19 | 12 | 10
Not Completed | 1 | 0 | 1 | 2
Period: Infusion 2
Arm/Group | MDD: Ketamine, Then Placebo | MDD: Placebo, Then Ketamine | Healthy Volunteers: Ketamine, Then Placebo | Healthy Volunteers:Placebo, Then Ketamine
Started | 19 | 18 | 11 | 11
Completed | 19 | 18 | 11 | 10
Not Completed | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Healthy Volunteer: Healthy volunteer patients
- Major Depressive Disorder (MDD): Patients diagnosed with Major Depressive Disorder (MDD)
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteer | Major Depressive Disorder (MDD) | Total
Number analyzed (Participants) | 25 | 42 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 41 | 66
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 25 | 41
  Male | 9 | 17 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 21 | 39 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 16 | 36 | 52
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: MADRS Score - Baseline
Description: Antidepressant effects were assessed using the Montgomery-Åsberg Depression Rating Scale (MADRS). It is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.
Time Frame: Baseline
Population: The analyses included subjects who were given Ketamine or Placebo.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ketamine - Healthy Volunteers; Placebo - Healthy Volunteers: Ketamine and placebo infusions were administered two weeks apart, with Ketamine's dose being 0.5 mg/kg to healthy volunteer patients
- Ketamine - MDD Patients; Placebo - MDD Patients: Ketamine and placebo infusions were administered two weeks apart, with Ketamine's dose being 0.5 mg/kg to patients with Major Depressive Disorders (MDD)
Arm/Group | Ketamine - Healthy Volunteers | Placebo - Healthy Volunteers | Ketamine - MDD Patients | Placebo - MDD Patients
Number analyzed (Participants) | 24 | 23 | 41 | 38
units on a scale | 1.17 (1.37) | 1.48 (1.78) | 33.83 (4.23) | 31.82 (5.84)

2. Primary Outcome: MADRS Score - Day 1 Following Intervention
Description: as for outcome 1
Time Frame: Day 1
Population: The analyses included subjects who were given Ketamine or Placebo.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine - Healthy Volunteers | Placebo - Healthy Volunteers | Ketamine - MDD Patients | Placebo - MDD Patients
Number analyzed (Participants) | 22 | 21 | 40 | 38
units on a scale | 2.45 (3.79) | 0.67 (1.15) | 23.73 (10.32) | 30.68 (5.50)

ADVERSE EVENTS:
Time Frame: 28 days
Groups:
- Healthy Volunteer: Ketamine; MDD: Ketamine: Ketamine and placebo infusions were administered two weeks apart, with Ketamine's dose being 0.5 mg/kg.
- Healthy Volunteer: Placebo; MDD: Placebo: Placebo and Ketamine infusions were administered two weeks apart, with Ketamine's dose being 0.5 mg/kg
Arm/Group | Healthy Volunteer: Ketamine | MDD: Ketamine | Healthy Volunteer: Placebo | MDD: Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/41 | 0/23 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/41 | 0/23 | 0/38
Other Adverse Events (participants affected / at risk) | 24/24 | 36/41 | 8/23 | 16/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Volunteer: Ketamine (N=24) | MDD: Ketamine (N=41) | Healthy Volunteer: Placebo (N=23) | MDD: Placebo (N=38)
Dizziness (Cardiac disorders) | 19 | 27 | 1 | 0
Dyspnoea (Cardiac disorders) | 0 | 2 | 0 | 0
Auditory disorder (Ear and labyrinth disorders) | 6 | 7 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 1 | 4 | 0 | 0
Vision blurred (Eye disorders) | 5 | 11 | 0 | 0
Visual impairment (Eye disorders) | 14 | 20 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 6 | 5 | 0 | 0
Dysgeusia (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 4 | 0 | 0
Oropharyngeal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Decreased appetite (General disorders) | 4 | 5 | 0 | 1
Energy increased (General disorders) | 2 | 3 | 0 | 0
Fatigue (General disorders) | 7 | 2 | 1 | 0
Feeling abnormal (General disorders) | 20 | 32 | 1 | 0
Flushing (General disorders) | 2 | 7 | 0 | 0
Hyperhidrosis (General disorders) | 1 | 3 | 0 | 0
Increased appetite (General disorders) | 0 | 2 | 0 | 1
Irritability (General disorders) | 0 | 2 | 0 | 1
Oedema (General disorders) | 0 | 0 | 1 | 0
Thirst (General disorders) | 1 | 0 | 0 | 0
Body temperature decreased (Investigations) | 2 | 6 | 0 | 1
Body temperature increased (Investigations) | 4 | 7 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2 | 1
Abnormal dreams (Nervous system disorders) | 1 | 2 | 0 | 0
Amnesia (Nervous system disorders) | 3 | 5 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Confusional state (Nervous system disorders) | 6 | 17 | 0 | 0
Disturbance in attention (Nervous system disorders) | 15 | 3 | 1 | 0
Dysarthria (Nervous system disorders) | 3 | 4 | 0 | 0
Headache (Nervous system disorders) | 2 | 4 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 14 | 24 | 1 | 0
Hypokinesia (Nervous system disorders) | 6 | 2 | 0 | 1
Insomnia (Nervous system disorders) | 5 | 7 | 2 | 5
Paraesthesia (Nervous system disorders) | 6 | 9 | 1 | 0
Parosmia (Nervous system disorders) | 0 | 2 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0 | 0 | 0
Sedation (Nervous system disorders) | 8 | 7 | 0 | 3
Slow speech (Nervous system disorders) | 6 | 17 | 0 | 0
Speech disorder (Nervous system disorders) | 11 | 20 | 0 | 0
Terminal insomnia (Nervous system disorders) | 0 | 1 | 0 | 2
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Vibratory sense increased (Nervous system disorders) | 1 | 5 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Dissociation (Psychiatric disorders) | 12 | 19 | 0 | 0
Euphoric mood (Psychiatric disorders) | 4 | 7 | 0 | 0
Fear (Psychiatric disorders) | 1 | 5 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 2 | 0 | 0
Libido decreased (Psychiatric disorders) | 1 | 0 | 0 | 0
Premenstrual syndrome (Psychiatric disorders) | 0 | 1 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 2 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 3 | 6 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT00088699/Prot_SAP_000.pdf